CLINICAL TRIAL: NCT06088212
Title: Reducing Cognitive Impairment by Management of Heart Failure as a Modifiable Risk Factor: the Cog-HF Trial
Brief Title: Reducing Cognitive Impairment by Management of Heart Failure as a Modifiable Risk Factor
Acronym: Cog-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P8510
Record Dates: First submitted 2023-09-27; First posted 2023-10-18 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure; Cognitive Impairment; Dementia; Left Ventricular Dysfunction; Cognitive Change; Cognitive Decline
MeSH Terms: conditions — Heart Failure; Cognitive Dysfunction; Dementia; Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Usual care patients will continue with the hospital follow-up plan and routine preventive care after hospital discharge.
- Intervention (Experimental): Intervention patients will receive a disease management program in addition to the usual care.
  Interventions: Other: Disease management program

INTERVENTIONS:
Other: Disease management program — The components of our DMP include:
  1. Intensive post-discharge education
  2. Home surveillance of signs and symptoms will be reviewed (weekly in the first month and monthly thereafter) in a telehealth consultation with patient and/or carer.
  3. Medical treatment involves a planned up-titration of cardioprotective medications that will proceed in the absence of advice from the general practitioner (GP) to the contrary. Close observation and frequent appointments are organised by the nurse with the patient's GP during up-titration period.
  4. Exercise program delivered by an exercise physiologist
  5. Maintenance phase of the DMP: During this maintenance phase, Intervention patients should have been fully transitioned to home care where they are managed by their GP at optimal doses of their medications. Repeated education and exercise guidance will continue with the carer, supported by our cardiac nurse and exercise physiologist via telehealth consultation bimonthly.
  Arms: Intervention

SUMMARY:
This study will test the feasibility and effectiveness of an innovative model of care for cognitively impaired patients with heart failure. This program aims to improve cognition, reduce dementia risk and cardiovascular events, and will be supported by innovative digital technology for wide scale rollout and implementation. Findings from this research will transform the way healthcare is delivered to cognitively impaired patients with heart disease who have a very high risk of developing dementia.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalised with HF as primary or secondary diagnosis.
2. At least mild cognitive impairment (CI) based on Montreal Cognitive Assessment (MoCA) on hospital discharge.

Exclusion Criteria:

1. Unable to provide written consent; requiring palliative care; or participating in another RCT
2. Recovery of cognitive function shortly after hospital discharge: to ensure that we only include patients with "true" CI, any patients with a repeated MoCA>25 at 2 weeks post-discharge will be excluded.
3. Terminal illness (eg. cancer) that may influence 12-month prognosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in MOCA score | 12 months
  Greater Montreal Cognitive Assessment (MOCA) score (ranging 0-30) is better

SECONDARY OUTCOMES:
Change in cardiac function | 12 months
  Cardiac function will be measured by echocardiography. Left ventricular global longitudinal strain will be the primary measure of cardiac function.
Change in 6-minute walk distance | 12 and 24 months
  Functional capacity will be based on 6-minute walk test
Change in quality of life | 12 and 24 months
  Quality of life specific to heart failure symptoms will be measured using a disease-specific quality of life questionnaire: Kansas City Cardiomyopathy Questionnaire
Change in MOCA score | 24 months
  Greater Montreal Cognitive Assessment (MOCA) score (ranging 0-30) is better
Change in brain volume via MRI measurement | 24 months
Change in hand grip strength | 12 and 24 months
Change in heart failure classification | 12 and 24 months
  Based on New York Heart Association classification

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Marwick, MBBS PhD MPH, Principal Investigator — Baker Heart and Diabetes Institute
Locations (1):
- Menzies Institute for Medical Research, Hobart, Tasmania, Australia

IPD SHARING:
Plan to Share IPD: No